CLINICAL TRIAL: NCT00415610
Title: Antihypertensive Treatment in Acute Cerebral Hemorrhage (ATACH)
Brief Title: Antihypertensive Treatment in Acute Cerebral Hemorrhage
Acronym: ATACH
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0609M93128; R01NS044976-01A2 (NIH)
Record Dates: First submitted 2006-12-21; First posted 2006-12-25 (Estimated); Results first posted 2015-09-07 (Estimated); Last update posted 2017-11-21 (Actual); Status verified 2017-11

CONDITIONS: Intracerebral Hemorrhage; Hypertension; Stroke
Keywords: cerebral hemorrhage; intracerebral hemorrhage; stroke; hypertension; blood pressure; nicardipine; antihypertensive agent; hematoma expansion
MeSH Terms: conditions — Cerebral Hemorrhage; Hypertension; Stroke | interventions — Nicardipine

STUDY DESIGN:
Intervention Model Description: Staged intensity levels of rapid intravenous antihypertensive control for elevated SBP in patients with intracerebral hemorrhage were implemented in 3 sequential treatment arms to assess the feasibility and tolerability (safety) of this treatment.
Masking Description: Open treatment assignment was employed because it is not safe to conceal SBP measurement. Patient data routinely entered by clinical staff were used to evaluate safety.
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Tier 1 (Other): Dose escalation:
  The scientists will investigate the potential consequences of controlling blood pressure with intravenous nicardipine to a range between 170 to 200 mmHg. Treatment with nicardipine must begin within 6 hours of symptom onset and will continue for an estimated 18 - 24 hours, until SBP is stabilized. The assigned SBP range will be maintained for 24 hours. After 24 hours, management of blood pressure is at the discretion of the primary physician.
  Interventions: Drug: nicardipine
- Tier 2 (Other): Dose escalation:
  The scientists will investigate the potential consequences of controlling blood pressure with intravenous nicardipine to a range between 140 to 170 mmHg. Treatment with nicardipine must begin within 6 hours of symptom onset and will continue for an estimated 18 - 24 hours, until SBP is stabilized. The assigned SBP range will be maintained for 24 hours. After 24 hours, management of blood pressure is at the discretion of the primary physician.
  Interventions: Drug: nicardipine
- Tier 3 (Other): Dose escalation:
  The scientists will investigate the potential consequences of controlling blood pressure with intravenous nicardipine to a range between 110 to 140 mmHg. Treatment with nicardipine must begin within 6 hours of symptom onset and will continue for an estimated 18 - 24 hours, until SBP is stabilized. The assigned SBP range will be maintained for 24 hours. After 24 hours, management of blood pressure is at the discretion of the primary physician.
  Interventions: Drug: nicardipine

INTERVENTIONS:
Drug: nicardipine — Intravenous (IV) nicardipine infusion. It is expected that the treatment duration will vary between 18 and 24 hours.
  * Started at 5mg/h
  * Titrated by 2.5mg/hour every 15 minutes to bring systolic blood pressure in target range for the applicable Tier. Max dose 15mg/hour *Once target systolic blood pressure reached, dose decreased by 2.5mg/hour every 15 minutes until systolic blood pressure maintained in the target range or the medication is discontinued.
  Other Names: Cardene, nicardipine hydrochloride

SUMMARY:
The purpose of this trial is to evaluate the safety and effectiveness of lowering blood pressure using nicardipine in persons with acute hypertension associated with intracerebral hemorrhage.

DETAILED DESCRIPTION:
An estimated 37,000 to 52,400 people in the United States have intracerebral hemorrhage (ICH) every year. ICH--a form of stroke that has poor outcome and is difficult to treat--is associated with the highest mortality rate of all strokes. Hematoma expansion has been identified as the most common cause of neurological deterioration in persons with ICH. Early evidence suggests that acute hypertension (HTN)-or elevated blood pressure-may make some individuals more susceptible to hematoma expansion. Treating HTN acutely may prevent hematoma expansion, however, the effect of aggressive HTN treatment has not been determined.

The purpose of this trial is to evaluate the treatment feasibility and safety of lowering blood pressure using nicardipine--an antihypertensive medication--in persons who have acute HTN associated with ICH.

This pilot study will enroll 60 individuals who qualify with a presenting systolic blood pressure of at least 170 mmHg, have an ICH, and can be evaluated and treatment initiated within 6 hours of onset of stroke symptoms. In a stepwise fashion, the scientists will investigate the potential consequences of controlling blood pressure with intravenous nicardipine at 3 sequential levels: 170 to 200 mmHg, 140 to 170 mmHg, and 110 to 140 mmHg. Twenty participants will be enrolled per level.

Treatment will last 18 to 24 hours. Participants will stay in the hospital for about 7 days (including 24 hours in the intensive care unit for close monitoring) and will return for 1-hour follow-up visits at 30 days and at 90 days after discharge from the hospital. During these visits participants will receive neurological assessments to determine their functional outcome. For participants, the study will be completed after the 90-day follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

* Age older than 18 years.
* Onset of new neurological signs of a stroke within 12 hours of the time to evaluation AND initiation of treatment with intravenous nicardipine.
* Clinical signs consistent with the diagnosis of stroke, including impairment of language, motor function, cognition, and/or gaze, vision, or neglect.
* The total GCS score is greater than 8 at the time of enrollment.
* CT scan demonstrates intraparenchymal hematoma with manual hematoma volume measurement less than 60 cc.
* ICH is supratentorial and is located in lobar, basal ganglionic, or thalamic based on the initial CT scan appearance.
* Admission systolic blood pressure greater than 170 mm Hg on two repeat measurements at least 5 minutes apart.
* Evidence of chronic hypertension.
* Subject is not considered a surgical candidate by the neurosurgery service.

Exclusion Criteria:

* Time of symptom onset cannot be reliably assessed.
* Previously known neoplasms, arteriovenous malformation, or aneurysms.
* Intracerebral hematoma considered to be related to trauma by the neurologist or neurosurgeon.
* ICH is located in the cortex or infratentorial regions such as pons or cerebellum.
* Blood is visualized in the subarachnoid space.
* Intravenous nicardipine cannot be initiated within 12 hours of symptom onset.
* Use of clonidine hydrochloride and other central alpha-agonist within the last 48 hours that have the potential of withdrawal hypertension.
* Pregnancy, lactation, or parturition within previous 30 days.
* Any history of bleeding diathesis or coagulopathy, including the use of warfarin.
* Use of heparin in the previous 48 hours and a prolonged partial thromboplastin time.
* Known atrial-ventricular heart block other than first degree, or sick sinus syndrome without a pacemaker.
* Intolerance to calcium channel blockers.
* Exposure to study medication in the preceding 24 hours prior to enrollment.
* A platelet counts less than 100 000/mm3.
* Major surgery within the previous six weeks.
* History of any intracranial hemorrhage (including intracerebral or subarachnoid hemorrhage) or hemorrhagic stroke.
* Seizure at onset of stroke.
* Blood glucose less than 50 mg/dL or greater than 400 mg/dL.
* Current participation in another research drug treatment protocol.
* Isolated ventricular blood on CT scan.
* Subject has a living will that precludes aggressive intensive care unit management.
* Subject has acute myocardial infarction or renal failure that precludes use of aggressive antihypertensive therapy.
* Subjects with unstable angina or acute myocardial infarction within 2 weeks prior to ICH.
* Subjects with renal insufficiency with serum creatinine greater than 2.0 mg/dl or on renal dialysis.
* Sinus tachycardia exceeding 120 beats per minute or supraventricular tachycardia is observed during initial evaluation.
* Ischemic stroke within 4 weeks of presentation.
* Congestive heart failure graded as class III and IV by New York Heart Association (NYHA) classification.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2005-07; Primary Completion 2007-09 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adnan I. Qureshi, MD, Principal Investigator — University of Minnesota
Locations (12):
- United States (12):
  - University of Southern California, Los Angeles, California
  - Kansas University Medical Center, Kansas City, Kansas
  - The University of Kansas School of Medicine, Wichita Via Christi Regional Medical Center, Kansas City, Kansas
  - Massachusetts General/Brigham Women's Hospital, Boston, Massachusetts
  - Clinical Coordinating Center: University of Minnesota, Fairview Hospital, Minneapolis, Minnesota
  - Saint Louis University, St Louis, Missouri
  - JFK Medical Center, Edison, New Jersey
  - University of Medicine and Dentistry of New Jersey, Newark, New Jersey
  - Columbia University Medical Center, New York, New York
  - Case Western Reserve University, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - Statistical Coordinating Center: Medical University of South Carolina, Charleston, South Carolina

IPD SHARING:
Plan to Share IPD: Undecided
consult investigator for options

REFERENCES:
- [Background] Qureshi AI. Antihypertensive Treatment of Acute Cerebral Hemorrhage (ATACH): rationale and design. Neurocrit Care. 2007;6(1):56-66. doi: 10.1385/ncc:6:1:56. PMID 17356194
- [Result] Qureshi AI, Palesch YY, Martin R, Novitzke J, Cruz-Flores S, Ehtisham A, Ezzeddine MA, Goldstein JN, Hussein HM, Suri MF, Tariq N; Antihypertensive Treatment of Acute Cerebral Hemorrhage Study Investigators. Effect of systolic blood pressure reduction on hematoma expansion, perihematomal edema, and 3-month outcome among patients with intracerebral hemorrhage: results from the antihypertensive treatment of acute cerebral hemorrhage study. Arch Neurol. 2010 May;67(5):570-6. doi: 10.1001/archneurol.2010.61. PMID 20457956
- [Result] Antihypertensive Treatment of Acute Cerebral Hemorrhage (ATACH) investigators. Antihypertensive treatment of acute cerebral hemorrhage. Crit Care Med. 2010 Feb;38(2):637-48. doi: 10.1097/CCM.0b013e3181b9e1a5. PMID 19770736
- [Result] Qureshi AI. Acute hypertensive response in patients with stroke: pathophysiology and management. Circulation. 2008 Jul 8;118(2):176-87. doi: 10.1161/CIRCULATIONAHA.107.723874. No abstract available. PMID 18606927
- [Result] Qureshi AI, Palesch YY, Martin R, Novitzke J, Cruz Flores S, Ehtisham A, Goldstein JN, Kirmani JF, Hussein HM, Suri MF, Tariq N; Antihypertensive Treatment of Acute Cerebral Hemorrhage Investigators. Systolic blood pressure reduction and risk of acute renal injury in patients with intracerebral hemorrhage. Am J Med. 2012 Jul;125(7):718.e1-6. doi: 10.1016/j.amjmed.2011.09.031. Epub 2012 May 4. PMID 22560810
- [Result] Qureshi AI, Palesch YY. Antihypertensive Treatment of Acute Cerebral Hemorrhage (ATACH) II: design, methods, and rationale. Neurocrit Care. 2011 Dec;15(3):559-76. doi: 10.1007/s12028-011-9538-3. PMID 21626077
- [Derived] Hussein HM, Tariq NA, Palesch YY, Qureshi AI; ATACH Investigators. Reliability of hematoma volume measurement at local sites in a multicenter acute intracerebral hemorrhage clinical trial. Stroke. 2013 Jan;44(1):237-9. doi: 10.1161/STROKEAHA.112.667220. Epub 2012 Dec 11. PMID 23233387

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients 18 years and older presenting to site hospital ED and ICU areas within 6 hours of symptom onset for ≤ 60 cc volume intracerebral hemorrhage, with GCS ≥ 8, systolic blood pressure ≥ 170 mmHg and meeting all inclusion/exclusion criteria were enrolled following consent by themselves or a family member/legally authorized representative.
Pre-assignment Details: A progressive, three-tiered approach to lowering systolic blood pressure with DSMB review after enrollment in each successive SBP range was completed. Safety was determined at each level before progressing to the next. Subjects meeting criteria and consenting to participate were considered enrolled and have been included in the data analysis.
Groups:
- Tier 1: Dose escalation: Initial range
  The scientists will investigate the potential consequences of controlling blood pressure with intravenous nicardipine at 170 to 200 mmHg
  Nicardipine: Intravenous (IV) nicardipine infusion. It is expected that the treatment duration will vary between 18 and 24 hours.
  * Started at 5mg/h
  * Titrated by 2.5mg/hour every 15 minutes to bring systolic blood pressure in target range for the applicable Tier. Max dose 15mg/hour *Once target systolic blood pressure reached, dose decreased by 2.5mg/hour every 15 minutes until systolic blood pressure maintained in the target range or the medication is discontinued.
  The DSMB will review safety, tolerability, and feasibility before escalation to the next level.
- Tier 2: Dose escalation:
  The scientists will investigate the potential consequences of controlling blood pressure with intravenous nicardipine at 140 to 170 mmHg
  Nicardipine: Intravenous (IV) nicardipine infusion. It is expected that the treatment duration will vary between 18 and 24 hours.
  * Started at 5mg/h
  * Titrated by 2.5mg/hour every 15 minutes to bring systolic blood pressure in target range for the applicable Tier. Max dose 15mg/hour *Once target systolic blood pressure reached, dose decreased by 2.5mg/hour every 15 minutes until systolic blood pressure maintained in the target range or the medication is discontinued.
  The DSMB will review safety, tolerability, and feasibility before escalation to the next level.
- Tier 3: Dose escalation:
  The scientists will investigate the potential consequences of controlling blood pressure with intravenous nicardipine at 110 to 140 mmHg
  Nicardipine: Intravenous (IV) nicardipine infusion. It is expected that the treatment duration will vary between 18 and 24 hours.
  * Started at 5mg/h
  * Titrated by 2.5mg/hour every 15 minutes to bring systolic blood pressure in target range for the applicable Tier. Max dose 15mg/hour *Once target systolic blood pressure reached, dose decreased by 2.5mg/hour every 15 minutes until systolic blood pressure maintained in the target range or the medication is discontinued.
Period: Overall Study
Arm/Group | Tier 1 | Tier 2 | Tier 3
Started | 18 | 20 | 22
Completed | 15 | 18 | 17
Not Completed | 3 | 2 | 5
Not completed — Death | 3 | 2 | 5

BASELINE CHARACTERISTICS:
Population: Group numbers were adjusted as adequate safety parameters were met in each successive treatment tier. A larger number of subjects were therefore evaluated in the final tier where safety is of greatest concern and SBP parameter is also of greatest challenge to meet.
Groups:
- Tier 1: Dose escalation:
  The scientists will investigate the potential consequences of controlling blood pressure with intravenous nicardipine to a range between 170 to 200 mmHg. Treatment with nicardipine must begin within 6 hours of symptom onset and will continue for an estimated 18 - 24 hours, until SBP is stabilized. The assigned SBP range will be maintained for 24 hours. After 24 hours, management of blood pressure is at the discretion of the primary physician.
  nicardipine: Intravenous (IV) nicardipine infusion. It is expected that the treatment duration will vary between 18 and 24 hours.
  * Started at 5mg/h
  * Titrated by 2.5mg/hour every 15 minutes to bring systolic blood pressure in target range for the applicable Tier. Max dose 15mg/hour *Once target systolic blood pressure reached, dose decreased by 2.5mg/hour every 15 minutes until systolic blood pressure maintained in the target range or the medication is discontinued.
- Tier 2: Dose escalation:
  The scientists will investigate the potential consequences of controlling blood pressure with intravenous nicardipine to a range between 140 to 170 mmHg. Treatment with nicardipine must begin within 6 hours of symptom onset and will continue for an estimated 18 - 24 hours, until SBP is stabilized. The assigned SBP range will be maintained for 24 hours. After 24 hours, management of blood pressure is at the discretion of the primary physician.
  nicardipine: Intravenous (IV) nicardipine infusion. It is expected that the treatment duration will vary between 18 and 24 hours.
  * Started at 5mg/h
  * Titrated by 2.5mg/hour every 15 minutes to bring systolic blood pressure in target range for the applicable Tier. Max dose 15mg/hour *Once target systolic blood pressure reached, dose decreased by 2.5mg/hour every 15 minutes until systolic blood pressure maintained in the target range or the medication is discontinued.
- Tier 3: Dose escalation:
  The scientists will investigate the potential consequences of controlling blood pressure with intravenous nicardipine to a range between 110 to 140 mmHg. Treatment with nicardipine must begin within 6 hours of symptom onset and will continue for an estimated 18 - 24 hours, until SBP is stabilized. The assigned SBP range will be maintained for 24 hours. After 24 hours, management of blood pressure is at the discretion of the primary physician.
  nicardipine: Intravenous (IV) nicardipine infusion. It is expected that the treatment duration will vary between 18 and 24 hours.
  * Started at 5mg/h
  * Titrated by 2.5mg/hour every 15 minutes to bring systolic blood pressure in target range for the applicable Tier. Max dose 15mg/hour *Once target systolic blood pressure reached, dose decreased by 2.5mg/hour every 15 minutes until systolic blood pressure maintained in the target range or the medication is discontinued.
- Total: Total of all reporting groups
Arm/Group | Tier 1 | Tier 2 | Tier 3 | Total
Number analyzed (Participants) | 18 | 20 | 22 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 62 (17.7) | 58.5 (13.0) | 65.1 (14.6) | 62 (15.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 8 | 9 | 26
  Male | 9 | 12 | 13 | 34
Race/Ethnicity, Customized [Number; unit: participants]
  White | 5 | 13 | 13 | 31
  Black | 11 | 7 | 7 | 25
  Others | 2 | 0 | 2 | 4
Region of Enrollment [Number; unit: participants]
  United States | 18 | 20 | 22 | 60
Baseline Measures - Timing of Treatment [Mean (Standard Deviation); unit: hours] — as mean time in hours from symptom onset
  hours
    Symptom onset to emergency department arrival | 1.72 (1.27) | 1.70 (1.13) | 1.86 (1.78) | 1.72 (1.37)
    Symptom onset to treatment initiation | 3.94 (1.45) | 4.13 (1.50) | 4.44 (2.08) | 4.19 (1.71)
Initial SBP [Median (Full Range); unit: millimeters of mercury (mmHg)] — as measured on ED arrival by automated cuff inflation device
  millimeters of mercury (mmHg) | 209 [178 to 255] | 212 [190 to 275] | 201 [171 to 300] | 208 [171 to 300]
Initial Hematoma Volume [Mean (Standard Deviation); unit: cubic centimeters] — as measured by central reader (vs. rapid ABC/2 method used for initial qualification), in cubic centimeters estimated total volume
  cubic centimeters | 15.45 (14.60) | 14.84 (17.15) | 10.94 (10.87) | 13.56 (14.24)
Baseline Measures of stroke symptom severity [Median (Full Range); unit: units on a scale] — As measured on ED arrival. The Glasgow Coma Scale (GCS) is most applicable in those critically ill and measures eye opening, verbal, and motor responses. Scores on the 3-component GCS may range from 3-15 and a lower score indicates a more severe condition. The National Institutes of Health Stroke Scale (NIHSS) is more sensitive for discerning subtle symptoms. Scores on the 11-component NIHSS may total between 0-42, with a higher score indicating a more severe stroke. ICH is an evolving condition and may worsen. NIHSS and GCS scores are used to measure changes in neurological status over time.
  units on a scale
    Initial NIHSS score | 11 [2 to 40] | 9 [0 to 25] | 8 [3 to 34] | 10 [0 to 40]
    Initial GCS | 14 [9 to 15] | 15 [8 to 15] | 15 [9 to 15] | 15 [8 to 15]
Duration of nicardipine infusion [Mean (Standard Deviation); unit: hours] — in total hours, as measured from initial start to final stop of any nicardipine administration
  hours | 12.93 (13.5) | 30.06 (23.8) | 45.82 (37.3) | 31.69 (30.75)
Maximum Dose of Nicardipine Used [Mean (Standard Deviation); unit: milligrams] — in total milligrams, as calculated by rate per hour by nicardipine volume % for total hours of infusion
  milligrams | 8.47 (5.75) | 8.90 (4.48) | 12.52 (6.76) | 10.10 (5.98)

OUTCOME MEASURES:

1. Primary Outcome: Particpants Who Achieve and Maintain the Systolic Blood Pressure Goals for Each Treatment Tier.
Description: Feasibility of treatment was assessed by whether SBP reduction and maintenance within the respective target range was achieved (treatment success) or not (treatment failure), and secondarily by whether a significant difference between treatment arms was achieved. Treatment failure was defined based on the observed hourly hourly minimum SBP remaining greater than the upper limit of the target range for 2 consecutive hours after initiation of nicardipine infusion. Spontaneous decline of SBP below the lower limit of the specific tier was not considered treatment failure as all such declines were asymptomatic.The lower number in the more intensive treatment groups reflects in part the greater challenge of rapidly lowering systolic blood pressure to a more intensive (lower) range, as a higher number of treatment failures as pre-defined by meeting the SBP range goal within 3 hours of symptom onset in this group predictably occurred.
Time Frame: Within 3 hours of symptom onset and sustained through 18-24 hours.
Population: All subjects were evaluated for achievement of the treatment goals.
Measure: Number; unit: participants
Arm/Group | Tier 1 | Tier 2 | Tier 3
Number analyzed (Participants) | 18 | 20 | 22
participants
  Meeting Criteria of initial SBP > 170 mmHg | 18 | 20 | 22
  Number treated within 3 hours of symptom onset | 7 | 5 | 6
  Treatment Failure, SBP not in range by 2 hours | 0 | 0 | 9
Statistical Analysis 1: Comparison: Tier 1 vs Tier 2 vs Tier 3; The hourly average (of maximum and minimum) SBP measurements were graphed with box-and-whiskers plot. In addition, a repeated measures analysis of the 25 average SBP (baseline and subsequent 24 hourly measures) was conducted with a mixed effects model (assuming autoregressive covariance structure in SAS version 9.1 PROC MIXED) to determine statistically the effect of treatment intensity (tier) on the average SBP over the 24 hrs with and without adjustment for baseline NIHSS score and age; Test type: Superiority or Other; p < 0.01, repeated measure — The repeated measure analysis of the hourly average SBP was calculated with and without adjusting for baseline NIHSS and age; Adjusted for initial deficit severity of using baseline NIHSS instead of GCS to better discriminate among patients with GCS score > 8

2. Primary Outcome: Number of Participants With Neurological Deteriorations (Decrease of 2 or More Points on the GCS Score or an Increase of 4 or More Points on the NIHSS Score) During the 24 Hour Treatment",
Description: Neurological status was monitored quantitatively and independently of other adverse events using two scales. The Glasgow Coma Scale (GCS) score measures level of consciousness in eye, motor, and verbal components. At least one point is given in each category. The scale ranges from 3 to 15, with 3 indicating deep unconsciousness and 15 indicating consciousness is not impaired. The National Institutes of Health Stroke Scale (NIHSS) quantifies neurologic deficits in 11 categories. Level of consciousness, horizontal eye movements, visual fields, facial palsy, movement in each limb, sensation, language and speech, and extinction or inattention on one side of the body are tested. Scores range from 0 to 42; 0 indicates normal function and higher scores indicate greater deficit severity.
Time Frame: within the first 72 hours of treatment initiation
Population: All subjects entered in the trial were followed and their data analyzed for safety measures. Not all subjects entered in the trial survived or remained in the trial to assess final outcomes at 1 or 3 months. When safety stopping rules could not have triggered after 18 initial subjects recruitment was adjusted to weight the subsequent tiers.
Measure: Number; unit: participants
Arm/Group | Tier 1 | Tier 2 | Tier 3
Number analyzed (Participants) | 18 | 20 | 22
participants | 1 | 2 | 4
Statistical Analysis 1: Comparison: Tier 1 vs Tier 2 vs Tier 3; Done as a surrogate to evaluate the relationship between early SBP reduction and safety events; Test type: Superiority or Other; p < .5, Wilcoxon rank sum test — Observed average SBP change at 2 hrs after treatment initiation between subjects who did or did not have neurologic deterioration within 24 hrs; Mean decrease measured for subjects with neurological deterioration and subjects without neurological deterioration

3. Primary Outcome: Total Number of Serious Adverse Events Within the Initial 72 Hours From Treatment Per Subject
Description: Serious adverse events were ascertained by site investigators using FDA-defined guidelines, defined as any untoward clinical events having been fatal, life-threatening, resulting in new or prolonged hospitalization, resulting in disability or congenital anomaly, or requiring intervention to prevent permanent impairment or damage. Subjects were followed closely from randomization through 90 days. The initial 72-hour period was chosen as the most meaningful time period for which to examine SAEs likely to be related to the acute safety of the study treatment.
Time Frame: from treatment initiation through 72 hours
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Tier 1 | Tier 2 | Tier 3
Number analyzed (Participants) | 18 | 20 | 22
Participants | 0 | 1 | 3

4. Secondary Outcome: Particpants Who Tolerate Rapid Systolic Blood Pressure Reduction and Maintain Treatment Goals
Description: The ability to maintain the Specified Systolic Blood Pressure Range for the 18-24 Hour Period without Neurological Deterioration or Side Effects
Time Frame: 3 months
Population: All subjects were analyzed by treatment arm for the presence of SAEs, neurological deterioration, symptomatic or asymptomatic hematoma expansion, and mortality in-hospital or within 3 months. Pre-specified safety stopping rules were used. The nature and relatedness of events was examined and overseen by an external Data safety and Monitoring Board.
Measure: Number; unit: participants
Arm/Group | Tier 1 | Tier 2 | Tier 3
Number analyzed (Participants) | 18 | 20 | 22
participants
  N with SAE within 72 hours | 0 | 1 | 3
  N with neurologic deterioration within 24 hours | 1 | 2 | 4
  N with symptomatic hematoma expansion | 0 | 1 | 4
  N with asymptomatic hematoma expansion | 6 | 2 | 3
  N with in-hospital mortality | 2 | 1 | 1
  N with 3-month mortality | 3 | 2 | 5
  N with 1-month favorable outcome, mRS 0-2 | 4 | 6 | 4
  N missing for 1-month outcome assessment | 3 | 3 | 2
  N with 3-month favorable outcome, mRS 0-2 | 8 | 9 | 7
  N missing for 3-month outcome assessment | 3 | 4 | 2

5. Other Pre Specified Outcome: Particpants Who Achieve Reduction of Blood Pressure and Maintain Treatment Goals (the Specified Systolic Blood Pressure Range for the 18-24 Hour Period) Without Neurological Deterioration or Side Effects Resulting in Death.
Description: The tolerability of the study treatment was further ascertained by examination of in-hospital, 1-month, or 3-month mortality in each treatment group.
  This pilot study was not powered (did not plan to enroll an adequate number of patients) to draw meaningful conclusions about individual adverse event categories, outcome measures, or to make comparisons between the treatment arms beyond the overall feasibility and tolerability of rapidly and significantly lowering SBP following intracerebral hemorrhage.
  The timing and magnitude of SBP reduction was also compared to the timing of individual safety events to further evaluate possible relationships between the study treatment, adverse events, and any recognizable safety concerns. This information is available in publication but is not able to be displayed on this website due to formatting restrictions.
Time Frame: From enrollment through 3 months
Population: Serious adverse events were monitored for all patients throughout the 3-month study period; when mortality resulted death was categorized as having occurred prior to or following hospital discharge. The 3-month mortality count includes deaths that occurred earlier. Survival was confirmed at hospital discharge, 1 month, and 3 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Tier 1 | Tier 2 | Tier 3
Number analyzed (Participants) | 18 | 20 | 22
Participants
  In-hospital mortality | 2 | 1 | 1
  Mortality at 3 months (also in participant flow) | 3 | 2 | 5
  Survival/no known death at 1 or 3 months (derived) | 13 | 17 | 16

ADVERSE EVENTS:
Time Frame: SAEs were collected from randomization through 90 +/- 14 days, but are reported through 72 hours (meaningful time in relation to treatment). Other AEs were collected through seven days from randomization or until hospital discharge, whichever came first.
Description: Safety stopping rules were established in the protocol based on the upper limit (by 95% confidence interval) for individual and cumulative rates of neurologic deterioration and serious adverse events (SAE) from previous studies in a manner similar to other phase I trials in acute stroke patents. Safety data was monitored by the NIH-appointed DSMB.
Arm/Group | Tier 1 | Tier 2 | Tier 3
Serious Adverse Events (participants affected / at risk) | 0/18 | 1/20 | 3/22
Other Adverse Events (participants affected / at risk) | 7/18 | 4/20 | 7/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tier 1 (N=18) | Tier 2 (N=20) | Tier 3 (N=22)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Acute respiratory distress syndrome (ARDS) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperglycemia and hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Symptomatic hematoma volume expansion (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) — defined as > 33 % increase in hematoma volume as measured by central reader between baseline and 24 hour head CT scans, accompanied by neurological deterioration or new neurological symptoms
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tier 1 (N=18) | Tier 2 (N=20) | Tier 3 (N=22)
Neurological deterioration within 24 hours (Nervous system disorders) | 1 (1) | 2 (2) | 4 (4) — defined as increase of 4 or more points on NIHSS or decrease of 2 or more points on GCS
Asymptomatic hematoma expansion (Nervous system disorders) | 6 (6) | 2 (2) | 3 (3) — Hematoma expansion is defined as > 33% increase in hematoma volume as measured by central reader between baseline and 24 hour head CT scans

LIMITATIONS AND CAVEATS:
Limited by small sample size and likelihood of imbalances in subject characteristics among the three tiers. Clinical measures may be insensitive. Not designed to provide comparative event rates and not powered toward prediction of clinical outcomes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No